CLINICAL TRIAL: NCT05026554
Title: Pathophysiological Characterization of Chronic Hand Eczema Subtypes and Atopic Dermatitis With Noninvasive Molecular and Imaging Techniques in Subjects With Moderate to Severe Chronic Hand Eczema, Subjects With Atopic Dermatitis, and Healthy Volunteers
Brief Title: Characterization of Chronic Hand Eczema
Status: Recruiting | Type: Observational
Sponsor: Dr. Robert Bissonnette (Other)
Responsible Party: Sponsor-Investigator, Dr. Robert Bissonnette, Principal Investigator, Innovaderm Research Inc.
Organization: Innovaderm Research Inc. (Other)
Other Study IDs: INNO-5024
Record Dates: First submitted 2021-08-05; First posted 2021-08-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Hand Eczema; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, skin tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- CHE: Adults with moderate to severe chronic hand eczema
  Interventions: Genetic: Tape stripping
- Healthy Volunteers: Healthy adults
  Interventions: Genetic: Tape stripping
- Atopic Dermatitis: subjects with moderate to severe AD
  Interventions: Genetic: Tape stripping

INTERVENTIONS:
Genetic: Tape stripping — Optional genetic analysis for chronic hand eczema

SUMMARY:
Prospective longitudinal study to characterize Choronic Hand Eczema (CHE) subtypes and Atopic Dermatitis (AD) with noninvasive molecular and imaging techniques, and assess changes through time and its association with quality of life.

DETAILED DESCRIPTION:
Prospective longitudinal study of adult patients with moderate to severe chronic hand eczema, subject with modreate to severe Atopic Dermatitis and healthy volenteers to assess changes in morphological parameters and molecular signatures with non-invasive techniques.In addition, disease severity and their association with occupation, smoking status, quality of life will be evaluated per CHE subtypes and compared to subjects with only AD. Samples and data collected from healthy volunteers will be used as controls in the analyses.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

1. Male or female subjects aged 18 to 65 years, inclusive, at the time of consent.
2. Subject is willing to participate and is capable of giving informed consent. Note: Consent must be obtained prior to any study-related procedures.
3. Subject must be willing to comply with all study procedures and must be available for the duration of the study.

   CHE subjects only:
4. Subject has at least a 6-month history of CHE before Screening (information obtained from medical chart or subject's physician, or directly from the subject).
5. Subject has moderate to severe CHE as defined by an IGA score of ≥3 at Screening and Day 1.
6. Subject has CHE covering ≥0.25% of BSA on palmar surface of hands at Screening and Day 1.
7. Subjects has CHE that can be categorized in one of the following CHE subtypes at Day 1:

   * Atopic hand eczema (without wet-work or excessive contact with irritants)
   * Irritant contact hand eczema without atopic disease
   * Hyperkeratotic hand eczema without atopic disease
   * Vesicular hand dermatitis without atopic disease
   * Allergic contact hand eczema without atopic disease
   * Idiopathic hand eczema without wet-work, excessive contact with irritants, atopic disease, hyperkeratotic morphology, allergic contact hand eczema and vesicular hand eczema.

   Subjects with only AD:
8. Subject has clinically confirmed diagnosis of active atopic dermatitis, according to Hanifin and Rajka criteria.
9. Subject has at least a 6-month history of AD and had no significant flares in AD for at least 4 weeks before Screening (information obtained from medical chart or subject's physician, or directly from the subject).
10. Subject has moderate to severe AD as defined by a vIGA-AD score of ≥3 at Screening and Day 1.
11. Subject has AD covering ≥0.5% of BSA at Screening and Day 1.
12. Subject has an AD lesion covering ≥0.25% of BSA on the forearm at Screening and Day 1.Healthy Volunteers only:
13. Subject is in good general health, according to the investigator's judgment based on medical history and physical examination.

Exclusion Criteria:

All subjects:

1. Subject has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the study assessments.
2. Subject has used systemic antibiotics within 2 weeks prior to Day 1.
3. Subject has used topical antibiotics within 1 week prior to Day 1.
4. Subject has used topical products containing urea or salicylic acid within 1 week prior to Day 1.
5. Subject has received any marketed or investigational biological agent within 12 weeks or 5 half-lives (whichever is longer) prior to Day 1.
6. Subject is currently receiving a nonbiological investigational product or device or has received one within 4 weeks prior to Day 1.
7. Subject has had excessive sun exposure, is planning a trip to a sunny climate, or has used tanning booths within 4 weeks prior to Day 1. Use of sunscreen products are recommended when exposure cannot be avoided.
8. Subject is a female who is pregnant or who is planning to become pregnant during the study.

   CHE subjects only:
9. Subject has clinically infected chronic hand eczema on hands and/or wrists.
10. Subject with suspected or proven hand eczema protein contact dermatitis.
11. Subject has used doxepin within 1 week prior to Day 1.
12. Subject has used hydroxyzine or diphenhydramine within 1 week prior to Day 1.
13. Subject has used any topical medicated treatment that could affect CHE within 1 week prior to Day 1, including, but not limited to, topical corticosteroids, topical retinoids, crisaborole, calcineurin inhibitors, tars, antimicrobials, medical devices, and bleach baths.
14. Subject has used alitretinoin, isotretinoin, acitretin or other systemic retinoids within 4 weeks before Day 1, or has not completely recovered from its side effects.
15. Subject has used systemic treatments (other than biologics) that could have an impact on CHE less than 4 weeks prior to Day 1 (eg, calcineurin inhibitors, methotrexate, cyclosporin, hydroxycarbamide [hydroxyurea], azathioprine), or systemic steroids (including oral or injectable corticosteroids).

    Note: Intranasal corticosteroids, eye or ear drops containing corticosteroids, and inhaled corticosteroids for stable medical conditions are allowed.
16. Subject has used dupilumab within 12 weeks prior to Day 1.
17. Subject has received any UV-B phototherapy (including tanning beds) or excimer laser within 4 weeks prior to Day 1.
18. Subject has had psoralen-UV-A (PUVA) treatment within 4 weeks prior to Day 1.

    Subjects with only AD:
19. Subject has clinically infected AD.
20. Subject has AD lesion on hand and/or feet at screening or Day 1.
21. Subject has received an intravenous immunoglobulin (IVIg) therapy within 12 weeks prior to Day 1.
22. Subject has used doxepin within 1 week prior to Day 1.
23. Subject has used hydroxyzine or diphenhydramine within 1 week prior to Day 1.
24. Subject has used any topical, medicated treatment that could affect AD within 1 week prior to Day 1, including, but not limited to, topical corticosteroids, crisaborole, calcineurin inhibitors, ruxolitinib, tars, antimicrobials, medical devices, and bleach baths.
25. Subject has used systemic treatments (other than biologics) that could affect AD less than 4 weeks prior to Day 1, including, but not limited to, retinoids, calcineurin inhibitors, methotrexate, cyclosporine, hydroxycarbamide (hydroxyurea), azathioprine, oral/injectable corticosteroids, baricitinib, upadacitinib, and abrocitinib.
26. Subject has used dupilumab within 12 weeks prior to Day 1.
27. Subject has received any UV-B phototherapy (including tanning beds) or excimer laser within 4 weeks prior to Day 1.
28. Subject has had PUVA treatment within 4 weeks prior to Day 1. Note: Intranasal corticosteroids and inhaled corticosteroids are allowed. Eye and ear drops containing corticosteroids are allowed.
29. Subject has used tralokinumab within 12 weeks prior to Day 1.

    Healthy Volunteers only:
30. Subject has history of atopic dermatitis, allergic rhinitis, or asthma.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 140 adult subjects will be enrolled in the study: 120 subjects with moderate to severe chronic hand eczema, and 20 healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2021-06-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Characterize differences in skin morphological parameters | 12 months
  Determine differences in skin morphological parameters between cohorts assessed with Hand Eczema Severity Index (HECSI). The HECSI scoring system incorporates both the extent and the intensity of the disease. Each hand will be divided into five areas (fingertips, fingers [except the tips], palms, back of hands and wrists). For each of these areas the intensity of the six following clinical signs: erythema, induration ⁄ papulation, vesicles, fissuring, scaling and oedema will be graded on the following scale: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe. For each location (total of both hands) the affected area will be given a score from 0 to 4 (0, 0%; 1, 1-25%; 2, 26-50%; 3, 51-75% and 4, 76-100%) for the extent of clinical symptoms.
Characterize differences in skin molecular signature | 12 months
  Determine differences in skin molecular signatures between cohorts by comparing gene expression profiles from skin tissue collected with tape strips.

SECONDARY OUTCOMES:
Determine disease severity impact on lifestyle | 12 months
  Evaluate correlation of lifestyle with disease severity. Lifestyle information will be captured with type of occupation performed daily by the subject. In addition, tobacco product usage will be collected with information on history (length of usage) and rate (the frequency of usage).
Determine disease severity impact on quality of life | 12 months
  Evaluate correlation of quality of life with disease severity. Quality of life will be captured with Dermatology Life Quality Index Questionnaire (DLQI). DLQI is a 10-item questionnaire used to measure the impact of skin disease on the quality of life of an affected person. Each item is scored from 0 to 3, giving a possible score range from 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
To biobank plasma, serum, whole blood, DNA (buffy coat), stool, skin surface material and skin tissue. | 10 years
  Blood and microbiome samples will be collected from all subjects. Blood samples will be collected for biomarker and gene expression analyses, and optional DNA analyses. Skin swab samples, and optional stool samples, will be collected for microbiome analyses, including bacterial load,diversity, and characterization. Collected samples not analyzed in them current study will be retained in a biobank for future research purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Bissonnette, MD, MSc, Principal Investigator — Innovaderm Research Inc.
Locations (1):
- Innovaderm Research, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No